CLINICAL TRIAL: NCT03349190
Title: A Retrospective, National, Multicenter Study Evaluating the Impact of Ulipristal Acetate (Esmya®) on Infertility to Infertile Women With Fibroids Managed With Assisted Reproduction Techniques (ART)
Brief Title: Impact of Esmya on Fertility to Infertile Women With Fibroids Managed With Assisted Reproduction Techniques
Acronym: NACRE
Status: Completed | Type: Observational
Sponsor: ASSOCIATION POUR LE DEVELOPPEMENT EN FECONDATION IN VITRO (Other)
Collaborators: Gedeon Richter Plc. (Industry)
Responsible Party: Principal Investigator, Catherine Rongieres, Head of the ART center of the University Hospital of Strasbourg, ASSOCIATION POUR LE DEVELOPPEMENT EN FECONDATION IN VITRO
Other Study IDs: 0001
Record Dates: First submitted 2017-11-10; First posted 2017-11-21 (Actual); Last update posted 2019-01-09 (Actual); Status verified 2019-01

CONDITIONS: Infertility, Female; Fibroid Uterus
MeSH Terms: conditions — Infertility, Female; Leiomyoma | interventions — ulipristal acetate

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: ULIPRISTAL ACETATE — Ulipristal Acetate (Esmya) administrated for fibroids indication before surgery and IVF/ICSI procedure(retrospective study)

SUMMARY:
Fibroid is a frequent pathology of infertile women. Its deleterious effect on the infertility would be due to the mechanical way.

The interest of the resection of intramural fibroids is discussed. It is necessary to measure the indication of a myomectomy, whatever the surgical procedure. On the one hand, it may cause important potential complications, and on the other hand, the surgery does not improve the parameters of the fertility.

Thus, it is a major stake to avoid the surgical operation. A decrease of the size of these fibroids by medical treatment is then a good option.

When the surgical treatment is necessary, a medical pre-surgical treatment is often proposed in order to decrease the symptomatology and to reduce the size of the fibroid to facilitate the surgery.

Acetate Ulipristal (UPA) has been marketed in this indication. Following the Pearl I-II studies, the first indication in France was a pre-surgical treatment for 3 months at a dose of 5 mg per day.

The Pearl III and IV studies evaluated the Esmya® administration as a long-term intermittent repeated treatment, giving to it a prominent position for the long-term management of symptomatic fibroids.

Furthermore, cases of pregnancy before surgery are frequently described in women with fibroids treated by UPA for a pre-IVF surgery.

5 to 10 % of women who are managed for infertility have fibroids and only 2% to 3% have this unique cause of infertility.

Then, some of patients followed in ART centers have been treated by UPA to reduce the fibroids size and/or to decrease the associate symptoms.

The aim of this study is to evaluate in the different French ART centers, the impact on fertilization of UPA administration for infertile women with fibroids and to describe the modalities of its prescriptions and to collect information regarding safety tolerance profile of Esmya® in this patient population.

DETAILED DESCRIPTION:
A retrospective, national, multicenter study

ELIGIBILITY:
Inclusion Criteria:

1. Age between 18 to 43 years 'old at the time of the beginning of ulipristal acetate intake
2. Women with fibroid at the time of ulipristal acetate prescription
3. Women with desire to have children and managed for infertility in an ART center (whatever the type of infertility treatment)
4. Women having received a treatment by ulipristal acetate
5. Data collected between 2013/12/01 and 2018/06/30 ; data collected between ulipristal acetate prescription until the term of pregnancy or embryo transfer failure (up to 4) or death/lost to follow up or ART treatment discontinuation

Exclusion Criteria:

none

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Infertile women with fibroids managed with assisted reproduction techniques (ART)
Sampling Method: Probability Sample
Enrollment: 127 (Actual)
Dates: Start 2017-12-29 (Actual); Primary Completion 2018-06-30 (Actual); Study Completion 2019-01-08 (Actual)

PRIMARY OUTCOMES:
Clinical pregnancy | 15 days
  Clinical pregnancy rate after maximum 4 embryos transferred by IVF/ICSI procedures ; pregnancy is defined by beta-hCG> 1000 or presence of a gestation sac

SECONDARY OUTCOMES:
Spontaneous pregnancy | at least 2 months
  Spontaneous pregnancy rate before first embryo transferred by IVF/ICSI procedures; pregnancy is defined by beta-hCG > 1000 or presence of a gestation sac
Live birth / miscarriage | 9 months
  Live birth rate / miscarriage rate
Fibroids size | Baseline (before ulipristal acetate administration) and 20 months
  Fibroids size reduction
Surgery rate | 3 months
  Rate of surgery
Surgery description | 3 months
  Description of the surgery type and surgery indication
Description of ulipristal acetate prescription | 20 months
  Reasons of the prescription, type of fibroids concerned, number of cycles of treatment, treatment duration
Safety impact on ulipristal acetate administration | 20 months
  Review of adverse drug reactions resulting in ulipristal acetate treatment modification or discontinuation
Ulipristal acetate safety analysis in infertile women with fibroids | 20 months
  Review of all serious adverse reactions (expected or unexpected) in this population

CONTACTS AND LOCATIONS:
Overall Officials: Catherine RONGIERES, MD, Principal Investigator — ADEFIV & University Hospitals of Strasbourg
Locations (23):
- France (22):
  - Chu Angers, Angers
  - Chu Besancon, Besançon
  - Chu Pellegrin, Bordeaux
  - Polyclinique Jean Villar, Bruges
  - Centre Hospitalier Intercommunal Creteil, Créteil
  - Chu Dijon, Dijon
  - Clinique Val D'Ouest, Écully
  - Chru Lille, Lille
  - Cpma Marseille, Marseille
  - Imr Rocca, Marseille
  - Chevalier, Montpellier
  - POUGET, Montpellier
  - CHU NICE, Nice
  - Chu Nimes, Nîmes
  - Ch Antoine Beclere, Paris
  - CH TENON, Paris
  - Maternite Bichat, Paris
  - MENARD, Paris
  - Port Royal - Chirurgie, Paris
  - Chu Rennes, Rennes
  - Cmco - University Hospitals of Strasbourg, Schiltigheim
  - Chu Toulouse, Toulouse
- Centre Hospitalier Territorial Gaston Bourret, Noumea, New Caledonia

IPD SHARING:
Plan to Share IPD: No